CLINICAL TRIAL: NCT01437059
Title: A Phase 1, Randomized, Single-blind, Placebo-Controlled, Single Ascending Dose, Safety, Tolerability and Pharmacokinetics Study of ALN-PCS02 in Subjects With Elevated LDL-Cholesterol (LDL-C)
Brief Title: Trial to Evaluate Safety and Tolerability of ALN-PCS02 in Subjects With Elevated LDL-Cholesterol (LDL-C)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALN-PCS02-001
Record Dates: First submitted 2011-09-19; First posted 2011-09-20 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Elevated LDL-Cholesterol (LDL-C)
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALN-PCS02 (Active Comparator)
  Interventions: Drug: ALN-PCS02
- Sterile Normal Saline (0.9% NaCl) (Placebo Comparator)
  Interventions: Drug: Sterile Normal Saline (0.9% NaCl)

INTERVENTIONS:
Drug: ALN-PCS02 — Dose levels between 15 and 400 μg/kg by intravenous (IV) infusion
  Arms: ALN-PCS02
Drug: Sterile Normal Saline (0.9% NaCl) — Calculated volume to match active comparator
  Arms: Sterile Normal Saline (0.9% NaCl)

SUMMARY:
The purpose of this study is to determine the safety, tolerability, pharmacokinetics and pharmacodynamics of a single dose of ALN-PCS02 in subjects with Elevated LDL-Cholesterol (LDL-C).

ELIGIBILITY:
Inclusion Criteria:

* Elevated LDL-C of >3.0 mmol/L and <5.7 mmol/L
* Fasting triglyceride concentration ≤2.8 mmol/L
* Body weight >60.0 kg; body mass index (BMI) between 19.00 kg/m2 and <35.00 kg/m2
* Adequate blood counts, liver and renal function
* May not received any lipid lowering drug/agent within the 30 days prior to the screening
* Non-smokers for at least 3 months
* Women of child-bearing potential must have a negative pregnancy test, cannot be breast feeding, and must use an adequate method of birth control
* Males agree to use appropriate contraception
* Willing and able to comply with protocol-required visit schedule and visit requirements and provide written informed consent

Exclusion Criteria:

* Known hepatitis B surface antigen (HBsAg), hepatitis B virus (HBV), hepatitis C virus (HCV) or human immunodeficiency virus (HIV) infection
* Multiple drug allergies or know sensitivity to oligonucleotide
* History of drug abuse and/or alcohol abuse
* Receiving an investigational agent within 3 months prior to study drug administration
* Subjects with safety laboratory test results deemed clinical significant by the Investigator;
* Received prescription drugs within 4 weeks of first dosing
* Subjects who have donated more than 500 mL of blood within the 3 months prior to ALN-PCS02 or placebo administration;
* Received megadose vitamin therapy or dietary supplements within 4 weeks prior to screening
* Subjects who have used prescription drugs within 4 weeks of first dosing
* Considered unfit for the study by the Principal Investigator
* Employee or family member of the sponsor or the clinical study site personnel

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects experiencing adverse events (AEs), serious adverse events (SAEs) and study drug discontinuation. | Up to 28 days

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ALN-PCS02 (Cmax, tmax, t1/2, AUC0-last, CL). | Up to 180 days
Effect of ALN-PCS02 on Circulating PCSK9 Levels (Determination of % Lowering of PCSK9 to pretreatment/Baseline PCSK9 Level). | Up to 28 days
Effect of ALN-PCS02 on Circulating LDL-c Levels (Determination of % Lowering of LDL-c to pretreatment/Baseline LDL-c Level). | Up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Amy Simon, MD, Study Director — Alnylam Pharmaceuticals
Locations (2):
- United Kingdom (2):
  - Clinical Site, Leeds
  - Clinical Site, London

REFERENCES:
- [Derived] Fitzgerald K, Frank-Kamenetsky M, Shulga-Morskaya S, Liebow A, Bettencourt BR, Sutherland JE, Hutabarat RM, Clausen VA, Karsten V, Cehelsky J, Nochur SV, Kotelianski V, Horton J, Mant T, Chiesa J, Ritter J, Munisamy M, Vaishnaw AK, Gollob JA, Simon A. Effect of an RNA interference drug on the synthesis of proprotein convertase subtilisin/kexin type 9 (PCSK9) and the concentration of serum LDL cholesterol in healthy volunteers: a randomised, single-blind, placebo-controlled, phase 1 trial. Lancet. 2014 Jan 4;383(9911):60-68. doi: 10.1016/S0140-6736(13)61914-5. Epub 2013 Oct 3. PMID 24094767